CLINICAL TRIAL: NCT01052636
Title: Intervention Program for Elderly Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Yea-Ing Lotus Shyu, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NHRI-EX90-9023PL; HMRPD9J10 (Other Grant/Funding Number: Chang Gung Memorial Hospital)
Record Dates: First submitted 2010-01-17; First posted 2010-01-20 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Hip Fracture
Keywords: Hip fracture; Intervention program; Elderly
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Patients receive only routine hospital care
- Experimental group (Experimental): Patients receive regular hospital routine care and interdisciplinary intervention program
  Interventions: Other: Interdisciplinary intervention program

INTERVENTIONS:
Other: Interdisciplinary intervention program — The intervention program developed for this study included three components: geriatric consultation service, rehabilitation program, and discharge-planning service.
  Arms: Experimental group

SUMMARY:
Specific Aims

The long-term objective of this study is to examine the effectiveness of an intervention program for older patients with hip fracture. First, an intervention program for elderly patients with hip fracture will be developed and implemented, then, the effectiveness of the intervention program will be examined. The specific aims are as follows:

1. To develop a well conceived and feasible protocol of hospital discharge and sub-acute care that involves the coordinated work of health care professionals (physicians, surgeons, nurses, and physical therapists) and the informal caregivers. The feasibility of implementing such a protocol within the context of an intervention study subject to the constraints of the clinical setting (i.e., CGMH) will be evaluated in a pilot study.
2. To conduct a randomized clinical trial to evaluate the outcomes and costs associated with the proposed hospital discharge/sub-acute care protocol for elderly patients with hip fracture. Both experimental and case study methods will be used. Information on outcome indicators including clinical outcomes, quality of life, self-care ability, family caregiving outcomes, patient and caregiver satisfaction, and services utilization will be collected and compared between the control group and the experimental group.
3. To conduct a validation clinical trial to verify the results of the primary randomized clinical trial and increase the generalization of the study findings.
4. To estimate the cost of this care model and its variations for individual patients.

DETAILED DESCRIPTION:
The percentage of elderly persons in Taiwan has continually increased, from 2.5% in 1951 to 8.26% in 1998; the current number of elderly is 1,811,335. As in other countries with an increasing aging population, hip fracture represents a major and growing health care problem in Taiwan. Hip fractures resulted in 15,000 hospital admissions in 1997. It is estimated that the incidence rate (per 100, 000) for hip fracture in Taiwan was 211 for Taiwan's elderly population in 1993, 10 times the incidence rate for the general population. Despite advanced treatments, the one-year mortality rate for hip fracture remains significant (15.4%), and a majority of patients never recover completely in terms of activities of daily living. The economic costs of hip fractures among the elderly are huge and families suffer from caregiving burdens. Many studies in the United States have shown that elderly patients with hip fracture can benefit from post-operative rehabilitation, early discharge planning, and transitional care. However, little is known about what interventions should be attempted for these patients and their family caregivers in Taiwan. The purpose of this experimental study is therefore to explore the effectiveness of an intervention program for older patients with hip fracture. The cost of this care model will also be estimated.

An intervention program will be developed in the first year. This program will be administered by a multidisciplinary health care team and will include a geriatric consultation service, an in-hospital and in-home rehabilitation program and a discharge planning component. During the first year, a pilot study consisting of 10 elderly patients with hip fracture and their caregivers in the experimental group and 10 in the control group will test the feasibility of the intervention program and establish a reference point for sample size modification. In the second and third years, a primary clinical trial will be conducted in Chang Gung Memorial Hospital in Lin Kuo. In this studies, 120 subjects who meet the sample criteria will be recruited and randomly assigned to the experimental and control group. Patients in the experimental group will receive regular hospital routine care and the intervention program. Patients in the control group will receive only routine hospital care. The outcome variables will include clinical outcomes, self-care ability, quality of life, family caregiving outcomes, patient and caregiver's satisfaction, and service utilization; data on those will be collected for one year after hospital discharge and compared between the experimental and control groups. Data on the cost of care will also be collected. A qualitative component will include in-depth interviews with five patients and their family caregivers from the experimental group, five from the control group and five health care providers, to explore the effects of the intervention program in detail. In the fourth and fifth years, a validation clinical trial will be conducted with 120 subjects. The intervention program will be implemented at a different medical center to validate the results of the primary clinical trial. The study results will provide suggestions for intervention protocols for elderly persons with hip fracture and guidelines for the development of intervention programs for other high-risk elderly persons in Taiwan. The findings also provide a reference for clinical and hospital administration decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Admitted from emergency room due to hip fracture
* Receiving hip arthroplasty or internal fixation
* Living in northern Taiwan

Exclusion Criteria:

* Severely cognitively impaired and completely unable to follow orders
* Terminally ill

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2001-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Quality of life | 1 year

SECONDARY OUTCOMES:
Clinical outcomes | 1 year
Self-care ability | 1 year
Family caregiving outcomes | 1 year
Patient and caregiver's satisfaction | 1 year
Service utilization | 1 year
Cost of care | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ing L Shyu, Ph.D., Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330
- [Derived] Shyu YI, Liang J, Wu CC, Cheng HS, Chen MC. An interdisciplinary intervention for older Taiwanese patients after surgery for hip fracture improves health-related quality of life. BMC Musculoskelet Disord. 2010 Sep 29;11:225. doi: 10.1186/1471-2474-11-225. PMID 20920220